CLINICAL TRIAL: NCT00562354
Title: A Phase 3, Open-Label Trial to Evaluate the Safety, Tolerability, and Immunogenicity of a 13vPnC When Administered to Healthy Japanese Adults Aged >= 65 Years and 50 to 64 Years in Japan Who Have Not Received a Previous Dose of 23-Valent Pneumococcal Polysaccharide Vaccine
Brief Title: Study Evaluating 13-valent Pneumococcal Conjugate Vaccine in Healthy Japanese Adults Aged >= 50 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6115A1-3004
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Results first posted 2011-11-11 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: Vaccines, Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Stratum 1: >= 65 years of age
  Interventions: Biological: 13vPnC
- 2 (Experimental): Stratum 2: 50 to 64 years of age
  Interventions: Biological: 13vPnC

INTERVENTIONS:
Biological: 13vPnC — 13vPnC for both stratum

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of the 13-valent pneumococcal conjugate (13vPnC) vaccine in healthy Japanese adults aged >= 50 years.

ELIGIBILITY:
Inclusion Criteria:

* Japanese descent male and female adults who do not have the potential to bear children >= 50 years of age.
* Determined to be eligible for the study based on medical history, physical examination, and clinical judgment. Subjects with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease 12 weeks before receipt of study vaccine, are eligible.
* Sexually active men must agree and commit to use a medically accepted form of contraception during the study and for at least 3 months after vaccination.

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine.
* Receipt of any vaccine within 30 days before study vaccination, except influenza vaccine.
* Documented S pneumoniae infection within the past 5 years before study vaccination.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (2):
- Japan (2):
  - Fukuoka, Fukuoka
  - Sumida-ku, Tokyo

REFERENCES:
- [Derived] Shiramoto M, Irie S, Juergens C, Yamaji M, Tamai S, Aizawa M, Belanger T, Gruber WC, Scott DA, Schmoele-Thoma B. Immunogenicity and safety of 13-valent pneumococcal conjugate vaccine when administered to healthy Japanese adults aged >/=50 years. An open-label trial. Hum Vaccin Immunother. 2014;10(7):1850-8. doi: 10.4161/hv.28633. PMID 25424792

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 271 participants were enrolled; 270 were vaccinated with study vaccine.
Groups:
- 13vPnC (50 to 64 Years of Age): 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a single dose of 0.5 milliliters (mL) intramuscularly (IM) to participants 50 to 64 years of age.
- 13vPnC (≥65 Years of Age): 13vPnC administered as a single dose of 0.5 mL IM to participants ≥65 years of age.
Period: Overall Study
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Started | 134 | 137
Received Study Treatment | 134 | 136
Evaluable Immunogenicity Population | 134 | 134
Completed | 134 | 135
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age) | Total
Number analyzed (Participants) | 134 | 134 | 268
Age Continuous [Mean (Standard Deviation); unit: years] | 57.5 (4.0) | 70.5 (4.4) | 64.0 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 70 | 146
  Male | 58 | 64 | 122

OUTCOME MEASURES:

1. Primary Outcome: Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for the 13 Serotypes 1 Month After Vaccination for Overall Population
Description: Serotype-specific antibody-mediated opsonophagocytic activity (functional antibodies) for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) as measured by a quantitative opsonophagocytic activity assay (OPA). OPA titers will be logarithmically transformed for analysis; geometric means calculated and expressed as geometric mean titers (GMTs). The 2-sided, 95% confidence intervals (CIs) on the GMTs were constructed by back transformation of the CIs for the mean of the logarithmically transformed assay results computed using the Student t distribution.
Time Frame: 1 month after vaccination
Population: Evaluable Immunogenicity population: treatments as randomized at all expected doses, blood drawn within specified timeframes, at least 1 valid and determinate assay result for proposed analysis, and no major protocol violations. N=number of participants with valid and determinate assay results for the specified serotype at both blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- 13vPnC Overall Population (50 to 64 and ≥65 Years of Age): 13vPnC administered as a single dose of 0.5 mL IM to participants 50 to 64 years of age and ≥65 years of age.
Arm/Group | 13vPnC Overall Population (50 to 64 and ≥65 Years of Age)
Number analyzed (Participants) | 263
titer
  Serotype 1 | 124 [101.5 to 150.7]
  Serotype 3 | 62 [53.1 to 73.4]
  Serotype 4 | 1333 [1054.4 to 1684.2]
  Serotype 5 | 215 [172.0 to 269.2]
  Serotype 6A | 2256 [1884.4 to 2700.3]
  Serotype 6B | 2861 [2406.4 to 3401.1]
  Serotype 7F | 1793 [1476.1 to 2177.7]
  Serotype 9V | 863 [652.9 to 1141.5]
  Serotype 14 | 1494 [1267.1 to 1761.9]
  Serotype 18C | 2082 [1683.5 to 2575.0]
  Serotype 19A | 874 [729.0 to 1047.8]
  Serotype 19F | 821 [655.7 to 1027.8]
  Serotype 23F | 538 [415.9 to 696.7]

2. Primary Outcome: Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for the 13 Serotypes 1 Month After Vaccination for Age Groups 50 to 64 Years and ≥65 Years
Description: Serotype-specific antibody-mediated opsonophagocytic activity (functional antibodies) for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) as measured by a quantitative opsonophagocytic activity assay (OPA). OPA titers will be logarithmically transformed for analysis; geometric means calculated and expressed as geometric mean titers (GMTs). The 2-sided, 95% CIs on the GMTs were constructed by back transformation of the CIs for the mean of the logarithmically transformed assay results computed using the Student t distribution.
Time Frame: 1 month after vaccination
Population: Evaluable Immunogenicity population. N=number of participants with valid and determinate assay results for the specified serotype at both blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Number analyzed (Participants) | 131 | 133
titer
  Serotype 1 | 93 [70.3 to 124.2] | 162 [124.0 to 212.6]
  Serotype 3 | 53 [42.0 to 67.8] | 73 [58.6 to 90.9]
  Serotype 4 | 1209 [830.1 to 1762.2] | 1464 [1098.8 to 1950.9]
  Serotype 5 | 159 [113.6 to 221.2] | 289 [214.7 to 387.9]
  Serotype 6A | 1667 [1283.1 to 2165.9] | 3082 [2431.0 to 3908.2]
  Serotype 6B | 2556 [1967.1 to 3320.8] | 3182 [2527.6 to 4004.7]
  Serotype 7F | 1469 [1075.6 to 2005.6] | 2218 [1772.6 to 2776.3]
  Serotype 9V | 738 [497.8 to 1094.8] | 1007 [675.2 to 1501.7]
  Serotype 14 | 1294 [1027.3 to 1629.2] | 1726 [1362.8 to 2185.2]
  Serotype 18C | 1503 [1087.0 to 2078.8] | 2862 [2187.0 to 3745.6]
  Serotype 19A | 616 [488.1 to 776.7] | 1241 [949.3 to 1621.7]
  Serotype 19F | 614 [438.9 to 858.0] | 1083 [804.7 to 1458.5]
  Serotype 23F | 361 [243.9 to 533.2] | 788 [566.6 to 1097.2]

3. Primary Outcome: Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rises (GMFRs) for the 13 Serotypes From Prevaccination to 1 Month After Vaccination for Overall Population
Description: Geometric mean fold rises (GMFRs) for the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from prevaccination to 1 month postvaccination were computed using the logarithmically transformed assay results. CI for the GMFRs are back transformations of a CI based on the Student t distribution for the logarithmically transformed assay results.
Time Frame: Prevaccination (Day 1), 1 month after vaccination
Population: Evaluable Immunogenicity population. N=number of participants with valid and determinate assay results for the specified serotype at both blood draws. GMFRs calculated using all participants with available data from both the prevaccination and postvaccination blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC Overall Population (50 to 64 and ≥65 Years of Age)
Number analyzed (Participants) | 263
fold rise
  Serotype 1 | 23.3 [19.17 to 28.31]
  Serotype 3 | 11.5 [9.69 to 13.67]
  Serotype 4 | 79.6 [55.79 to 113.47]
  Serotype 5 | 42.4 [33.64 to 53.51]
  Serotype 6A | 48.8 [35.04 to 67.87]
  Serotype 6B | 16.6 [11.79 to 23.51]
  Serotype 7F | 137.2 [99.26 to 189.69]
  Serotype 9V | 13.4 [9.17 to 19.46]
  Serotype 14 | 12.4 [9.23 to 16.76]
  Serotype 18C | 52.9 [38.41 to 72.82]
  Serotype 19A | 41.9 [32.46 to 54.22]
  Serotype 19F | 42.7 [32.34 to 56.25]
  Serotype 23F | 47.5 [35.23 to 63.92]

4. Primary Outcome: Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rises (GMFRs) for the 13 Serotypes From Prevaccination to 1 Month After Vaccination for Age Groups 50 to 64 Years and ≥65 Years
Description: as for outcome 3
Time Frame: Prevaccination (Day 1), 1 month after vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Number analyzed (Participants) | 131 | 133
fold rise
  Serotype 1 | 18.7 [14.02 to 24.91] | 28.8 [22.17 to 37.52]
  Serotype 3 | 9.8 [7.62 to 12.49] | 13.6 [10.66 to 17.24]
  Serotype 4 | 50.7 [29.40 to 87.32] | 123.3 [78.54 to 193.67]
  Serotype 5 | 34.3 [24.61 to 47.90] | 52.0 [37.59 to 71.88]
  Serotype 6A | 32.3 [20.50 to 50.81] | 74.7 [46.39 to 120.22]
  Serotype 6B | 11.2 [6.98 to 18.09] | 24.1 [14.68 to 39.60]
  Serotype 7F | 99.9 [62.24 to 160.40] | 192.5 [124.26 to 298.35]
  Serotype 9V | 7.3 [4.42 to 12.02] | 24.2 [14.02 to 41.86]
  Serotype 14 | 10.6 [7.00 to 16.08] | 14.6 [9.46 to 22.44]
  Serotype 18C | 31.0 [19.68 to 48.75] | 89.2 [57.54 to 138.25]
  Serotype 19A | 25.3 [18.75 to 34.13] | 69.5 [46.56 to 103.89]
  Serotype 19F | 25.3 [17.42 to 36.65] | 70.3 [47.39 to 104.14]
  Serotype 23F | 40.8 [26.53 to 62.89] | 54.7 [36.11 to 82.94]

5. Secondary Outcome: Comparison of Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for the 13 Serotypes 1 Month After Vaccination by Age Group
Description: as for outcome 2
Time Frame: 1 month after vaccination
Population: Evaluable Immunogenicity population. N=number of participants with determinate antibody titers for the specified serotype. GMTs calculated using all participants with available data for the specified blood draw.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Number analyzed (Participants) | 134 | 134
titer
  Serotype 1 | 93 [70.3 to 124.2] | 164 [125.1 to 213.9]
  Serotype 3 | 54 [42.2 to 67.9] | 73 [58.6 to 90.2]
  Serotype 4 | 1331 [967.6 to 1831.7] | 1786 [1390.9 to 2293.9]
  Serotype 5 | 171 [123.9 to 236.4] | 294 [219.9 to 393.0]
  Serotype 6A | 1663 [1287.0 to 2147.9] | 3148 [2502.2 to 3960.6]
  Serotype 6B | 2462 [1905.0 to 3181.7] | 3383 [2721.3 to 4204.8]
  Serotype 7F | 1484 [1097.7 to 2005.3] | 2247 [1818.6 to 2776.7]
  Serotype 9V | 797 [557.1 to 1138.9] | 1062 [735.5 to 1533.7]
  Serotype 14 | 1289 [1033.8 to 1608.1] | 1740 [1386.0 to 2183.8]
  Serotype 18C | 1530 [1114.5 to 2099.8] | 2922 [2243.8 to 3804.0]
  Serotype 19A | 604 [483.8 to 754.4] | 1267 [979.8 to 1637.9]
  Serotype 19F | 627 [454.7 to 863.7] | 1094 [814.1 to 1470.4]
  Serotype 23F | 398 [276.1 to 575.1] | 824 [596.3 to 1137.5]
Statistical Analysis 1: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 1: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of OPA GMTs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean titer = 0.6, 95% CI 2-sided [0.39 to 0.84] — Ratio of GMTs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 2: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 3: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of OPA GMTs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean titer = 0.7, 95% CI 2-sided [0.54 to 1.01] — Ratio of GMTs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 3: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 4: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of OPA GMTs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean titer = 0.7, 95% CI 2-sided [0.50 to 1.11] — Ratio of GMTs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 4: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 5: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of OPA GMTs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean titer = 0.6, 95% CI 2-sided [0.38 to 0.90] — Ratio of GMTs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 5: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 6A: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of OPA GMTs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean titer = 0.5, 95% CI 2-sided [0.37 to 0.74] — Ratio of GMTs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 6: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 6B: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of OPA GMTs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean titer = 0.7, 95% CI 2-sided [0.52 to 1.02] — Ratio of GMTs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 7: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 7F: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of OPA GMTs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean titer = 0.7, 95% CI 2-sided [0.46 to 0.95] — Ratio of GMTs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 8: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 9V: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of OPA GMTs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean titer = 0.7, 95% CI 2-sided [0.45 to 1.25] — Ratio of GMTs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 9: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 14: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of OPA GMTs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean titer = 0.7, 95% CI 2-sided [0.54 to 1.02] — Ratio of GMTs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 10: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 18C: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of OPA GMTs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean titer = 0.5, 95% CI 2-sided [0.35 to 0.79] — Ratio of GMTs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 11: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 19A: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of OPA GMTs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean titer = 0.5, 95% CI 2-sided [0.34 to 0.67] — Ratio of GMTs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 12: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 19F: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of OPA GMTs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean titer = 0.6, 95% CI 2-sided [0.37 to 0.88] — Confidence intervals for the ratio are back transformation of the CIs based on the Student t distribution for the mean difference of the logarithmically transformed assay results
Statistical Analysis 13: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 23F: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of OPA GMTs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean titer = 0.5, 95% CI 2-sided [0.30 to 0.79] — Ratio of GMTs were calculated by back transformation of the mean difference between age groups on the logarithmic scale

6. Secondary Outcome: Percentage of Participants Achieving Serotype Specific OPA Titers ≥ Lower Limit of Quantitation (LLOQ) for the 13 Serotypes 1 Month After Vaccination for Overall Population
Description: For OPA assays serotype-specific lower limit of quantitation (LLOQ) was derived the 13 serotypes: serotype 1=18; 3=12; 4=21; 5=29; 6A=37; 6B=43; 7F=210; 9V=345; 14=35; 18C=31; 19A=18; 19F=48; 23F=13. For each serotype the proportion (percentage of participants) achieving an OPA titer of at least 1:LLOQ was computed along with exact, 2-sided 95% confidence interval for the proportion.
Time Frame: 1 month after vaccination
Population: Evaluable Immunogenicity population. N=number of participants with determinate postvaccination OPA antibody titers to the given serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC Overall Population (50 to 64 and ≥65 Years of Age)
Number analyzed (Participants) | 266
percentage of participants
  Serotype 1 | 91.6 [87.6 to 94.7]
  Serotype 3 | 89.8 [85.6 to 93.2]
  Serotype 4 | 95.2 [91.8 to 97.5]
  Serotype 5 | 88.6 [84.0 to 92.2]
  Serotype 6A | 98.5 [96.2 to 99.6]
  Serotype 6B | 98.5 [96.2 to 99.6]
  Serotype 7F | 96.5 [93.5 to 98.4]
  Serotype 9V | 89.1 [84.7 to 92.5]
  Serotype 14 | 98.5 [96.2 to 99.6]
  Serotype 18C | 96.6 [93.7 to 98.4]
  Serotype 19A | 98.9 [96.7 to 99.8]
  Serotype 19F | 94.2 [90.6 to 96.7]
  Serotype 23F | 89.2 [84.8 to 92.7]

7. Secondary Outcome: Percentage of Participants Achieving Serotype Specific OPA Titers ≥ Lower Limit of Quantitation (LLOQ) for the 13 Serotypes 1 Month After Vaccination for Age Groups 50 to 64 Years and ≥65 Years
Description: as for outcome 6
Time Frame: 1 month after vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Number analyzed (Participants) | 133 | 134
percentage of participants
  Serotype 1 | 89.1 [82.5 to 93.9] | 94.0 [88.6 to 97.4]
  Serotype 3 | 87.9 [81.1 to 92.9] | 91.8 [85.8 to 95.8]
  Serotype 4 | 93.5 [87.6 to 97.2] | 96.9 [92.3 to 99.1]
  Serotype 5 | 85.8 [78.5 to 91.4] | 91.3 [85.0 to 95.6]
  Serotype 6A | 97.7 [93.5 to 99.5] | 99.2 [95.9 to 100.0]
  Serotype 6B | 97.7 [93.4 to 99.5] | 99.3 [95.9 to 100.0]
  Serotype 7F | 93.9 [88.4 to 97.3] | 99.2 [95.7 to 100.0]
  Serotype 9V | 88.6 [82.0 to 93.5] | 89.5 [83.0 to 94.1]
  Serotype 14 | 98.5 [94.6 to 99.8] | 98.5 [94.6 to 99.8]
  Serotype 18C | 95.5 [90.4 to 98.3] | 97.7 [93.5 to 99.5]
  Serotype 19A | 99.2 [95.8 to 100.0] | 98.5 [94.6 to 99.8]
  Serotype 19F | 93.0 [87.1 to 96.7] | 95.3 [90.2 to 98.3]
  Serotype 23F | 86.2 [79.0 to 91.6] | 92.3 [86.3 to 96.2]

8. Secondary Outcome: Comparison of Percentage of Participants Achieving Serotype Specific OPA Titers ≥ Lower Limit of Quantitation (LLOQ) for the 13 Serotypes 1 Month After Vaccination by Age Group
Description: as for outcome 6
Time Frame: 1 month after vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Number analyzed (Participants) | 133 | 134
percentage of participants
  Serotype 1 | 89.1 [82.5 to 93.9] | 94.0 [88.6 to 97.4]
  Serotype 3 | 87.9 [81.1 to 92.9] | 91.8 [85.8 to 95.8]
  Serotype 4 | 93.5 [87.6 to 97.2] | 96.9 [92.3 to 99.1]
  Serotype 5 | 85.8 [78.5 to 91.4] | 91.3 [85.0 to 95.6]
  Serotype 6A | 97.7 [93.5 to 99.5] | 99.2 [95.9 to 100.0]
  Serotype 6B | 97.7 [93.4 to 99.5] | 99.3 [95.9 to 100.0]
  Serotype 7F | 93.9 [88.4 to 97.3] | 99.2 [95.7 to 100.0]
  Serotype 9V | 88.6 [82.0 to 93.5] | 89.5 [83.0 to 94.1]
  Serotype 14 | 98.5 [94.6 to 99.8] | 98.5 [94.6 to 99.8]
  Serotype 18C | 95.5 [90.4 to 98.3] | 97.7 [93.5 to 99.5]
  Serotype 19A | 99.2 [95.8 to 100.0] | 98.5 [94.6 to 99.8]
  Serotype 19F | 93.0 [87.1 to 96.7] | 95.3 [90.2 to 98.3]
  Serotype 23F | 86.2 [79.0 to 91.6] | 92.3 [86.3 to 96.2]
Statistical Analysis 1: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 1: To assess differences between reporting groups exact, 2-sided 95% CIs on the difference in proportions between reporting groups were calculated (50 to 64 years age group minus ≥ 65 years age group); Test type: Superiority or Other; difference in proportions = -4.9, 95% CI 2-sided [-12.1 to 2.0]
Statistical Analysis 2: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 3: To assess differences between reporting groups exact, 2-sided 95% CIs on the difference in proportions between reporting groups were calculated (50 to 64 years age group minus ≥ 65 years age group); Test type: Superiority or Other; difference in proportions = -3.9, 95% CI 2-sided [-11.6 to 3.5]
Statistical Analysis 3: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 4: To assess differences between reporting groups exact, 2-sided 95% CIs on the difference in proportions between reporting groups were calculated (50 to 64 years age group minus ≥ 65 years age group); Test type: Superiority or Other; difference in proportions = -3.4, 95% CI 2-sided [-9.6 to 2.2]
Statistical Analysis 4: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 5: To assess differences between reporting groups exact, 2-sided 95% CIs on the difference in proportions between reporting groups were calculated (50 to 64 years age group minus ≥ 65 years age group); Test type: Superiority or Other; difference in proportions = -5.5, 95% CI 2-sided [-13.7 to 2.5]
Statistical Analysis 5: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 6A: To assess differences between reporting groups exact, 2-sided 95% CIs on the difference in proportions between reporting groups were calculated (50 to 64 years age group minus ≥ 65 years age group); Test type: Superiority or Other; difference in proportions = -1.5, 95% CI 2-sided [-5.7 to 2.1]
Statistical Analysis 6: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 6B: To assess differences between reporting groups exact, 2-sided 95% CIs on the difference in proportions between reporting groups were calculated (50 to 64 years age group minus ≥ 65 years age group); Test type: Superiority or Other; difference in proportions = -1.6, 95% CI 2-sided [-5.9 to 2.1]
Statistical Analysis 7: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 7F: To assess differences between reporting groups exact, 2-sided 95% CIs on the difference in proportions between reporting groups were calculated (50 to 64 years age group minus ≥ 65 years age group); Test type: Superiority or Other; difference in proportions = -5.3, 95% CI 2-sided [-10.8 to -0.9]
Statistical Analysis 8: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 9V: To assess differences between reporting groups exact, 2-sided 95% CIs on the difference in proportions between reporting groups were calculated (50 to 64 years age group minus ≥ 65 years age group); Test type: Superiority or Other; difference in proportions = -0.8, 95% CI 2-sided [-8.7 to 6.9]
Statistical Analysis 9: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 14: To assess differences between reporting groups exact, 2-sided 95% CIs on the difference in proportions between reporting groups were calculated (50 to 64 years age group minus ≥ 65 years age group); Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-4.0 to 4.1]
Statistical Analysis 10: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 18C: To assess differences between reporting groups exact, 2-sided 95% CIs on the difference in proportions between reporting groups were calculated (50 to 64 years age group minus ≥ 65 years age group); Test type: Superiority or Other; difference in proportions = -2.3, 95% CI 2-sided [-7.6 to 2.5]
Statistical Analysis 11: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 19A: To assess differences between reporting groups exact, 2-sided 95% CIs on the difference in proportions between reporting groups were calculated (50 to 64 years age group minus ≥ 65 years age group); Test type: Superiority or Other; difference in proportions = 0.8, 95% CI 2-sided [-2.8 to 4.7]
Statistical Analysis 12: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 19F: To assess differences between reporting groups exact, 2-sided 95% CIs on the difference in proportions between reporting groups were calculated (50 to 64 years age group minus ≥ 65 years age group); Test type: Superiority or Other; difference in proportions = -2.4, 95% CI 2-sided [-8.8 to 3.7]
Statistical Analysis 13: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 23F: To assess differences between reporting groups exact, 2-sided 95% CIs on the difference in proportions between reporting groups were calculated (50 to 64 years age group minus ≥ 65 years age group); Test type: Superiority or Other; difference in proportions = -6.2, 95% CI 2-sided [-14.1 to 1.5]

9. Secondary Outcome: Percentage of Participants Achieving ≥2-fold Rise in Serotype Specific OPA Titers for the 13 Serotypes 1 Month After Vaccination for Overall Population
Description: For each serotype the proportion (percentage of participants) achieving at least a 2-fold rise on the serotype-specific antibody titer from prevaccination to 1 month postvaccination was computed along with exact, 2-sided 95% confidence interval for the proportion.
Time Frame: 1 month after vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC Overall Population (50 to 64 and ≥65 Years of Age)
Number analyzed (Participants) | 263
percentage of participants
  Serotype 1 | 89.7 [85.4 to 93.1]
  Serotype 3 | 84.4 [79.5 to 88.6]
  Serotype 4 | 84.9 [79.2 to 89.5]
  Serotype 5 | 87.1 [82.2 to 91.1]
  Serotype 6A | 84.5 [79.5 to 88.8]
  Serotype 6B | 68.4 [62.0 to 74.2]
  Serotype 7F | 86.1 [81.1 to 90.2]
  Serotype 9V | 61.3 [54.8 to 67.6]
  Serotype 14 | 67.2 [61.0 to 73.0]
  Serotype 18C | 85.6 [80.7 to 89.7]
  Serotype 19A | 92.3 [88.3 to 95.3]
  Serotype 19F | 88.0 [83.3 to 91.8]
  Serotype 23F | 81.3 [75.9 to 86.0]

10. Secondary Outcome: Percentage of Participants Achieving ≥2-fold Rise in Serotype Specific OPA Titers for the 13 Serotypes 1 Month After Vaccination for Age Groups 50 to 64 Years and ≥65 Years
Description: as for outcome 9
Time Frame: 1 month after vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Number analyzed (Participants) | 131 | 133
percentage of participants
  Serotype 1 | 86.0 [78.8 to 91.5] | 93.2 [87.5 to 96.9]
  Serotype 3 | 81.7 [74.0 to 87.9] | 87.1 [80.2 to 92.3]
  Serotype 4 | 79.2 [70.0 to 86.6] | 90.4 [83.0 to 95.3]
  Serotype 5 | 84.7 [77.0 to 90.7] | 89.4 [82.6 to 94.3]
  Serotype 6A | 82.0 [74.3 to 88.3] | 87.1 [79.9 to 92.4]
  Serotype 6B | 61.7 [52.2 to 70.6] | 74.6 [65.9 to 82.0]
  Serotype 7F | 82.5 [74.8 to 88.7] | 89.8 [82.9 to 94.6]
  Serotype 9V | 52.5 [43.1 to 61.8] | 70.0 [61.0 to 78.0]
  Serotype 14 | 62.4 [53.3 to 70.9] | 72.0 [63.3 to 79.7]
  Serotype 18C | 80.3 [72.3 to 86.8] | 90.8 [84.4 to 95.1]
  Serotype 19A | 92.7 [86.7 to 96.6] | 91.9 [85.7 to 96.1]
  Serotype 19F | 86.1 [78.6 to 91.7] | 89.8 [83.3 to 94.5]
  Serotype 23F | 80.0 [71.7 to 86.7] | 82.5 [74.8 to 88.7]

11. Secondary Outcome: Comparison of Percentage of Participants Achieving ≥2-fold Rise in Serotype Specific OPA Titers for the 13 Serotypes 1 Month After Vaccination by Age Group
Description: as for outcome 9
Time Frame: 1 month after vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Number analyzed (Participants) | 131 | 133
percentage of participants
  Serotype 1 | 86.0 [78.8 to 91.5] | 93.2 [87.5 to 96.9]
  Serotype 3 | 81.7 [74.0 to 87.9] | 87.1 [80.2 to 92.3]
  Serotype 4 | 79.2 [70.0 to 86.6] | 90.4 [83.0 to 95.3]
  Serotype 5 | 84.7 [77.0 to 90.7] | 89.4 [82.6 to 94.3]
  Serotype 6A | 82.0 [74.3 to 88.3] | 87.1 [79.9 to 92.4]
  Serotype 6B | 61.7 [52.2 to 70.6] | 74.6 [65.9 to 82.0]
  Serotype 7F | 82.5 [74.8 to 88.7] | 89.8 [82.9 to 94.6]
  Serotype 9V | 52.5 [43.1 to 61.8] | 70.0 [61.0 to 78.0]
  Serotype 14 | 62.4 [53.3 to 70.9] | 72.0 [63.3 to 79.7]
  Serotype 18C | 80.3 [72.3 to 86.8] | 90.8 [84.4 to 95.1]
  Serotype 19A | 92.7 [86.7 to 96.6] | 91.9 [85.7 to 96.1]
  Serotype 19F | 86.1 [78.6 to 91.7] | 89.8 [83.3 to 94.5]
  Serotype 23F | 80.0 [71.7 to 86.7] | 82.5 [74.8 to 88.7]
Statistical Analysis 1: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; difference in proportions = -7.2, 95% CI 2-sided [-15.1 to 0.3]
Statistical Analysis 2: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; difference in proportions = -5.4, 95% CI 2-sided [-14.5 to 3.5]
Statistical Analysis 3: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; difference in proportions = -11.2, 95% CI 2-sided [-21.4 to -1.0]
Statistical Analysis 4: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; difference in proportions = -4.7, 95% CI 2-sided [-13.5 to 3.9]
Statistical Analysis 5: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 5]; Test type: Superiority or Other; difference in proportions = -5.1, 95% CI 2-sided [-14.3 to 4.0]
Statistical Analysis 6: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 6]; Test type: Superiority or Other; difference in proportions = -12.9, 95% CI 2-sided [-24.6 to -0.8]
Statistical Analysis 7: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; difference in proportions = -7.3, 95% CI 2-sided [-16.3 to 1.5]
Statistical Analysis 8: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 8]; Test type: Superiority or Other; difference in proportions = -17.5, 95% CI 2-sided [-29.5 to -5.0]
Statistical Analysis 9: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 9]; Test type: Superiority or Other; difference in proportions = -9.6, 95% CI 2-sided [-21.4 to 2.4]
Statistical Analysis 10: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; difference in proportions = -10.5, 95% CI 2-sided [-19.3 to -1.3]
Statistical Analysis 11: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 11]; Test type: Superiority or Other; difference in proportions = 0.8, 95% CI 2-sided [-6.2 to 7.9]
Statistical Analysis 12: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 12]; Test type: Superiority or Other; difference in proportions = -3.8, 95% CI 2-sided [-12.2 to 4.5]
Statistical Analysis 13: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; difference in proportions = -2.5, 95% CI 2-sided [-12.5 to 7.3]

12. Secondary Outcome: Percentage of Participants Achieving ≥4-fold Rise in Serotype Specific OPA Titers for the 13 Serotypes 1 Month After Vaccination for Overall Population
Description: For each serotype the proportion (percentage of participants) achieving at least a 4-fold rise on the serotype-specific antibody titer from prevaccination to 1 month postvaccination was computed along with exact, 2-sided 95% confidence interval for the proportion.
Time Frame: 1 month after vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC Overall Population (50 to 64 and ≥65 Years of Age)
Number analyzed (Participants) | 263
percentage of participants
  Serotype 1 | 88.9 [84.5 to 92.5]
  Serotype 3 | 76.0 [70.4 to 81.1]
  Serotype 4 | 74.6 [68.1 to 80.4]
  Serotype 5 | 85.1 [79.9 to 89.3]
  Serotype 6A | 75.4 [69.6 to 80.6]
  Serotype 6B | 57.0 [50.4 to 63.4]
  Serotype 7F | 81.6 [76.1 to 86.2]
  Serotype 9V | 50.0 [43.5 to 56.5]
  Serotype 14 | 56.0 [49.6 to 62.2]
  Serotype 18C | 77.0 [71.4 to 82.0]
  Serotype 19A | 85.9 [80.9 to 90.0]
  Serotype 19F | 78.8 [73.2 to 83.7]
  Serotype 23F | 75.6 [69.7 to 80.8]

13. Secondary Outcome: Percentage of Participants Achieving ≥4-fold Rise in Serotype Specific OPA Titers for the 13 Serotypes 1 Month After Vaccination for Age Groups 50 to 64 Years and ≥65 Years
Description: as for outcome 12
Time Frame: 1 month after vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Number analyzed (Participants) | 131 | 133
percentage of participants
  Serotype 1 | 86.0 [78.8 to 91.5] | 91.7 [85.7 to 95.8]
  Serotype 3 | 73.3 [64.8 to 80.6] | 78.8 [70.8 to 85.4]
  Serotype 4 | 65.3 [55.2 to 74.5] | 83.7 [75.1 to 90.2]
  Serotype 5 | 83.9 [76.0 to 90.0] | 86.2 [78.8 to 91.7]
  Serotype 6A | 69.5 [60.8 to 77.4] | 81.5 [73.5 to 87.9]
  Serotype 6B | 51.3 [41.8 to 60.7] | 62.3 [53.1 to 70.9]
  Serotype 7F | 77.0 [68.6 to 84.0] | 86.4 [78.9 to 92.0]
  Serotype 9V | 36.4 [27.8 to 45.8] | 63.3 [54.1 to 71.9]
  Serotype 14 | 52.8 [43.7 to 61.8] | 59.2 [50.1 to 67.9]
  Serotype 18C | 70.9 [62.1 to 78.6] | 83.1 [75.5 to 89.1]
  Serotype 19A | 85.5 [78.0 to 91.2] | 86.3 [79.0 to 91.8]
  Serotype 19F | 73.0 [64.2 to 80.6] | 84.4 [76.9 to 90.2]
  Serotype 23F | 71.7 [62.7 to 79.5] | 79.4 [71.2 to 86.1]

14. Secondary Outcome: Comparison of Percentage of Participants Achieving ≥4-fold Rise in Serotype Specific OPA Titers for the 13 Serotypes 1 Month After Vaccination by Age Group
Description: as for outcome 12
Time Frame: 1 month after vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Number analyzed (Participants) | 131 | 133
percentage of participants
  Serotype 1 | 86.0 [78.8 to 91.5] | 91.7 [85.7 to 95.8]
  Serotype 3 | 73.3 [64.8 to 80.6] | 78.8 [70.8 to 85.4]
  Serotype 4 | 65.3 [55.2 to 74.5] | 83.7 [75.1 to 90.2]
  Serotype 5 | 83.9 [76.0 to 90.0] | 86.2 [78.8 to 91.7]
  Serotype 6A | 69.5 [60.8 to 77.4] | 81.5 [73.5 to 87.9]
  Serotype 6B | 51.3 [41.8 to 60.7] | 62.3 [53.1 to 70.9]
  Serotype 7F | 77.0 [68.6 to 84.0] | 86.4 [78.9 to 92.0]
  Serotype 9V | 36.4 [27.8 to 45.8] | 63.3 [54.1 to 71.9]
  Serotype 14 | 52.8 [43.7 to 61.8] | 59.2 [50.1 to 67.9]
  Serotype 18C | 70.9 [62.1 to 78.6] | 83.1 [75.5 to 89.1]
  Serotype 19A | 85.5 [78.0 to 91.2] | 86.3 [79.0 to 91.8]
  Serotype 19F | 73.0 [64.2 to 80.6] | 84.4 [76.9 to 90.2]
  Serotype 23F | 71.7 [62.7 to 79.5] | 79.4 [71.2 to 86.1]
Statistical Analysis 1: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; difference in proportions = -5.7, 95% CI 2-sided [-13.8 to 2.1]
Statistical Analysis 2: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; difference in proportions = -5.5, 95% CI 2-sided [-15.9 to 5.0]
Statistical Analysis 3: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; difference in proportions = -18.3, 95% CI 2-sided [-30.1 to -5.9]
Statistical Analysis 4: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; difference in proportions = -2.3, 95% CI 2-sided [-11.6 to 6.9]
Statistical Analysis 5: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 5]; Test type: Superiority or Other; difference in proportions = -11.9, 95% CI 2-sided [-22.6 to -1.2]
Statistical Analysis 6: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 6]; Test type: Superiority or Other; difference in proportions = -11.0, 95% CI 2-sided [-23.8 to 1.9]
Statistical Analysis 7: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; difference in proportions = -9.5, 95% CI 2-sided [-19.3 to 0.4]
Statistical Analysis 8: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 8]; Test type: Superiority or Other; difference in proportions = -26.9, 95% CI 2-sided [-39.0 to -14.1]
Statistical Analysis 9: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 9]; Test type: Superiority or Other; difference in proportions = -6.4, 95% CI 2-sided [-18.7 to 6.1]
Statistical Analysis 10: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; difference in proportions = -12.2, 95% CI 2-sided [-22.6 to -1.7]
Statistical Analysis 11: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 11]; Test type: Superiority or Other; difference in proportions = -0.8, 95% CI 2-sided [-9.8 to 8.1]
Statistical Analysis 12: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 12]; Test type: Superiority or Other; difference in proportions = -11.4, 95% CI 2-sided [-21.7 to -1.2]
Statistical Analysis 13: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; difference in proportions = -7.7, 95% CI 2-sided [-18.5 to 3.4]

15. Secondary Outcome: Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for the 13 Serotypes 1 Month After Vaccination for Overall Population
Description: Serotype-specific IgG antibody concentrations for the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F), as measured by enzyme-linked immunosorbent assay (ELISA). IgG concentrations will be logarithmically transformed for analysis; geometric means calculated and expressed as geometric mean concentration (GMC) in micrograms per mL (mcg/mL). The 2-sided, 95% CIs on the GMCs were constructed by back transformation of the CIs for the mean of the logarithmically transformed assay results computed using the Student t distribution.
Time Frame: 1 month after vaccination
Population: Evaluable Immunogenicity population. N=number of participants with valid and determinate assay results for the specified serotype at both blood draws. GMCs calculated using all participants with available data for both the specified blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC Overall Population (50 to 64 and ≥65 Years of Age)
Number analyzed (Participants) | 268
mcg/mL
  Serotype 1 | 6.05 [5.05 to 7.24]
  Serotype 3 | 1.53 [1.36 to 1.72]
  Serotype 4 | 4.57 [3.87 to 5.39]
  Serotype 5 | 8.34 [7.28 to 9.56]
  Serotype 6A | 7.93 [6.79 to 9.25]
  Serotype 6B | 8.31 [7.08 to 9.75]
  Serotype 7F | 10.36 [9.01 to 11.91]
  Serotype 9V | 9.62 [8.29 to 11.16]
  Serotype 14 | 19.23 [16.47 to 22.44]
  Serotype 18C | 13.90 [12.10 to 15.96]
  Serotype 19A | 19.13 [16.54 to 22.13]
  Serotype 19F | 7.77 [6.40 to 9.43]
  Serotype 23F | 12.23 [10.34 to 14.46]

16. Secondary Outcome: Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for the 13 Serotypes 1 Month After Vaccination for Age Groups 50 to 64 Years and ≥65 Years
Description: as for outcome 15
Time Frame: 1 month after vaccination
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Number analyzed (Participants) | 134 | 134
mcg/mL
  Serotype 1 | 4.65 [3.65 to 5.91] | 7.95 [6.11 to 10.35]
  Serotype 3 | 1.38 [1.17 to 1.62] | 1.69 [1.43 to 2.00]
  Serotype 4 | 3.63 [2.88 to 4.59] | 5.78 [4.58 to 7.28]
  Serotype 5 | 6.74 [5.62 to 8.09] | 10.32 [8.46 to 12.60]
  Serotype 6A | 6.72 [5.48 to 8.24] | 9.37 [7.44 to 11.80]
  Serotype 6B | 6.71 [5.42 to 8.32] | 10.28 [8.12 to 13.00]
  Serotype 7F | 8.90 [7.34 to 10.80] | 12.10 [9.90 to 14.80]
  Serotype 9V | 6.55 [5.32 to 8.05] | 14.22 [11.72 to 17.25]
  Serotype 14 | 16.73 [13.59 to 20.59] | 22.12 [17.59 to 27.83]
  Serotype 18C | 10.47 [8.62 to 12.70] | 18.53 [15.35 to 22.37]
  Serotype 19A | 13.51 [11.16 to 16.36] | 27.09 [22.07 to 33.25]
  Serotype 19F | 4.99 [3.92 to 6.37] | 11.92 [8.98 to 15.82]
  Serotype 23F | 9.38 [7.35 to 11.98] | 15.93 [12.75 to 19.91]

17. Secondary Outcome: Comparison of Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for the 13 Serotypes 1 Month After Vaccination by Age Group
Description: as for outcome 15
Time Frame: 1 month after vaccination
Population: Evaluable Immunogenicity population. N=number of participants with determinate antibody concentration for the specified serotype. GMCs calculated using all participants with available data for the specified blood draw.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Number analyzed (Participants) | 134 | 134
mcg/mL
  Serotype 1 | 4.65 [3.65 to 5.91] | 7.69 [5.94 to 9.96]
  Serotype 3 | 1.35 [1.15 to 1.58] | 1.69 [1.43 to 2.00]
  Serotype 4 | 3.53 [2.80 to 4.45] | 5.35 [4.25 to 6.75]
  Serotype 5 | 6.74 [5.62 to 8.09] | 10.32 [8.46 to 12.60]
  Serotype 6A | 6.72 [5.48 to 8.24] | 9.45 [7.51 to 11.89]
  Serotype 6B | 6.71 [5.42 to 8.32] | 10.28 [8.12 to 13.00]
  Serotype 7F | 8.90 [7.34 to 10.80] | 12.09 [9.92 to 14.73]
  Serotype 9V | 6.55 [5.32 to 8.05] | 14.22 [11.72 to 17.25]
  Serotype 14 | 16.73 [13.59 to 20.59] | 22.13 [17.63 to 27.80]
  Serotype 18C | 10.47 [8.62 to 12.70] | 18.48 [15.32 to 22.28]
  Serotype 19A | 13.51 [11.16 to 16.36] | 27.09 [22.07 to 33.25]
  Serotype 19F | 4.69 [3.72 to 5.91] | 11.21 [8.51 to 14.77]
  Serotype 23F | 9.38 [7.35 to 11.98] | 15.93 [12.75 to 19.91]
Statistical Analysis 1: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 1: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of IgG GMCs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean concentration = 0.60, 95% CI 2-sided [0.43 to 0.86] — Ratio of GMCs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 2: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 3: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of IgG GMCs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean concentration = 0.80, 95% CI 2-sided [0.63 to 1.00] — Ratio of GMCs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 3: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 4: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of IgG GMCs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean concentration = 0.66, 95% CI 2-sided [0.48 to 0.91] — Ratio of GMCs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 4: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 5: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of IgG GMCs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean concentration = 0.65, 95% CI 2-sided [0.50 to 0.85] — Ratio of GMCs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 5: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 6A: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of IgG GMCs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean concentration = 0.71, 95% CI 2-sided [0.52 to 0.97] — Ratio of GMCs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 6: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 6B: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of IgG GMCs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean concentration = 0.65, 95% CI 2-sided [0.48 to 0.90] — Ratio of GMCs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 7: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 7F: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of IgG GMCs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean concentration = 0.74, 95% CI 2-sided [0.56 to 0.97] — Ratio of GMCs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 8: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 9V: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of IgG GMCs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean concentration = 0.46, 95% CI 2-sided [0.35 to 0.61] — Ratio of GMCs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 9: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 14: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of IgG GMCs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean concentration = 0.76, 95% CI 2-sided [0.56 to 1.03] — Ratio of GMCs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 10: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 18C: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of IgG GMCs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean concentration = 0.57, 95% CI 2-sided [0.43 to 0.74] — Ratio of GMCs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 11: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 19A: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of IgG GMCs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean concentration = 0.50, 95% CI 2-sided [0.38 to 0.66] — Ratio of GMCs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 12: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 19F: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of IgG GMCs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean concentration = 0.42, 95% CI 2-sided [0.29 to 0.60] — Ratio of GMCs were calculated by back transformation of the mean difference between age groups on the logarithmic scale
Statistical Analysis 13: Comparison: 13vPnC (50 to 64 Years of Age) vs 13vPnC (≥65 Years of Age); Serotype 23F: To assess differences between reporting groups, 2-sided 95% CIs for the ratio of IgG GMCs were constructed by back transformation of the CIs for the mean difference of the log-transformed assay results computed using the Student t-distribution; Test type: Superiority or Other; ratio of geometric mean concentration = 0.59, 95% CI 2-sided [0.42 to 0.82] — Ratio of GMCs were calculated by back transformation of the mean difference between age groups on the logarithmic scale

18. Secondary Outcome: Immunoglobulin G (IgG) Geometric Mean Fold Rises (GMFRs) for the 13 Serotypes 1 Month After Vaccination for Overall Population
Description: as for outcome 3
Time Frame: 1 month after vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC Overall Population (50 to 64 and ≥65 Years of Age)
Number analyzed (Participants) | 268
fold rise
  Serotype 1 | 11.38 [9.65 to 13.43]
  Serotype 3 | 2.89 [2.60 to 3.22]
  Serotype 4 | 15.89 [13.45 to 18.77]
  Serotype 5 | 4.15 [3.64 to 4.74]
  Serotype 6A | 4.23 [3.69 to 4.84]
  Serotype 6B | 4.32 [3.76 to 4.96]
  Serotype 7F | 11.59 [9.96 to 13.49]
  Serotype 9V | 8.56 [7.43 to 9.87]
  Serotype 14 | 6.79 [5.78 to 7.98]
  Serotype 18C | 12.94 [11.01 to 15.21]
  Serotype 19A | 7.36 [6.39 to 8.48]
  Serotype 19F | 6.03 [5.10 to 7.14]
  Serotype 23F | 7.80 [6.70 to 9.07]

19. Secondary Outcome: Immunoglobulin G (IgG) Geometric Mean Fold Rises (GMFRs) for the 13 Serotypes 1 Month After Vaccination for Age Groups 50 to 64 Years and ≥65 Years
Description: as for outcome 3
Time Frame: 1 month after vaccination
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Number analyzed (Participants) | 134 | 134
fold rise
  Serotype 1 | 8.86 [7.08 to 11.09] | 14.77 [11.65 to 18.72]
  Serotype 3 | 2.40 [2.07 to 2.79] | 3.47 [2.98 to 4.05]
  Serotype 4 | 11.33 [9.06 to 14.19] | 22.44 [17.75 to 28.38]
  Serotype 5 | 3.23 [2.70 to 3.85] | 5.34 [4.42 to 6.46]
  Serotype 6A | 3.32 [2.80 to 3.94] | 5.39 [4.38 to 6.64]
  Serotype 6B | 3.26 [2.72 to 3.92] | 5.71 [4.68 to 6.97]
  Serotype 7F | 9.10 [7.39 to 11.22] | 14.88 [12.00 to 18.45]
  Serotype 9V | 5.76 [4.77 to 6.95] | 12.80 [10.56 to 15.51]
  Serotype 14 | 5.93 [4.78 to 7.35] | 7.80 [6.13 to 9.91]
  Serotype 18C | 9.92 [7.99 to 12.31] | 16.96 [13.42 to 21.43]
  Serotype 19A | 5.12 [4.30 to 6.10] | 10.57 [8.60 to 12.99]
  Serotype 19F | 3.80 [3.07 to 4.71] | 9.43 [7.45 to 11.94]
  Serotype 23F | 6.26 [5.02 to 7.80] | 9.71 [7.91 to 11.91]

20. Secondary Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination for Overall Population
Description: Local reactions reported using electronic diary. Redness and swelling scaled as Any (redness or swelling present); Mild (2.5 centimeters [cm] to 5.0 cm); Moderate (5.1 to 10.0 cm); Severe (> 10.0 cm). Pain as Any (pain present); Mild (awareness of symptom, easily tolerated); Moderate (discomfort enough to cause interference with usual activity); Severe (incapacitating, inability to do usual activity). Limitation of arm movement scaled as Any (limitation present); Mild (some limitation); Moderate (unable to move above head, able to move above shoulder); Severe (unable to move above shoulder).
Time Frame: Day 1 through 14
Population: Safety population included all participants who received the study treatment. N=number of participants with analyzable data for reactogenicity events. Participants may be represented in more than 1 category.
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Overall Population (50 to 64 and ≥65 Years of Age)
Number analyzed (Participants) | 238
percentage of participants
  Redness: any | 14.4
  Redness: mild | 8.7
  Redness: moderate | 9.3
  Redness: severe | 0.5
  Swelling: any | 11.5
  Swelling: mild | 7.2
  Swelling: moderate | 5.8
  Swelling: severe | 0.5
  Pain: any | 48.3
  Pain: mild | 46.1
  Pain: moderate | 9.6
  Pain: severe | 0.5
  Limitation of arm movement: any | 53.2
  Limitation of arm movement: mild | 52.2
  Limitation of arm movement: moderate | 4.4
  Limitation of arm movement: severe | 1.5

21. Secondary Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 14 Days After Vaccination for Age Groups 50 to 64 Years and ≥65 Years
Description: as for outcome 20
Time Frame: Day 1 through 14
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Groups:
- 13vPnC (50 to 64 Years of Age): 13vPnC administered as a single dose of 0.5 mL IM to participants 50 to 64 years of age.
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Number analyzed (Participants) | 120 | 118
percentage of participants
  Redness: any | 7.1 | 20.9
  Redness: mild | 7.1 | 10.0
  Redness: moderate | 1.0 | 16.7
  Redness: severe | 0.0 | 0.9
  Swelling: any | 8.1 | 14.7
  Swelling: mild | 7.1 | 7.3
  Swelling: moderate | 2.0 | 9.3
  Swelling: severe | 0.0 | 0.9
  Pain: any | 52.2 | 44.3
  Pain: mild | 49.6 | 42.6
  Pain: moderate | 8.9 | 10.3
  Pain: severe | 1.0 | 0.0
  Limitation of arm movement: any | 53.0 | 53.4
  Limitation of arm movement: mild | 51.8 | 52.5
  Limitation of arm movement: moderate | 5.1 | 3.7
  Limitation of arm movement: severe | 2.1 | 0.9

22. Secondary Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination for Overall Population
Description: Systemic events reported using electronic diary. Fever scaled as Any (≥37.5 degrees Celsius [C]); Mild (≥37.5 but <38.5 degrees C); Moderate (≥38.5 but <39 degrees C); Severe (≥39 to ≤40 degrees C); Potentially life-threatening (>40 degrees C). Other systemic events include Fatigue, Headache, Chills, Rash, Vomiting, Decreased appetite, New muscle pain, Any aggravated muscle pain, New joint pain, and Any aggravated joint pain.
Time Frame: Day 1 through 14
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC Overall Population (50 to 64 and ≥65 Years of Age)
Number analyzed (Participants) | 228
percentage of participants
  Fever: any ≥37.5 degrees C | 3.4
  Fever: mild ≥37.5 but <38.5 degrees C | 2.9
  Fever: moderate ≥38.5 but <39 degrees C | 0.5
  Fatigue | 31.2
  Headache | 19.9
  Chills | 12.7
  Rash | 10.7
  Vomiting | 2.0
  Decreased appetite | 12.6
  New muscle pain | 31.8
  Any aggravated muscle pain | 10.1
  New joint pain | 11.0
  Any aggravated joint pain | 6.3

23. Secondary Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 14 Days After Vaccination for Age Groups 50 to 64 Years and ≥65 Years
Description: as for outcome 22
Time Frame: Day 1 through 14
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Number analyzed (Participants) | 112 | 116
percentage of participants
  Fever any ≥37.5 degrees C | 3.1 | 3.7
  Fever: mild ≥37.5 but <38.5 degrees C | 2.0 | 3.7
  Fever: moderate ≥38.5 but <39 degrees C | 1.0 | 0.0
  Fatigue | 38.8 | 24.1
  Headache | 26.0 | 14.4
  Chills | 14.9 | 10.8
  Rash | 8.2 | 13.1
  Vomiting | 3.1 | 0.9
  Decreased appetite | 16.2 | 9.3
  New muscle pain | 34.3 | 29.5
  Any aggravated muscle pain | 11.2 | 9.1
  New joint pain | 10.0 | 11.8
  Any aggravated joint pain | 7.1 | 5.5

ADVERSE EVENTS:
Time Frame: Adverse events reported via the electronic-diary were collected within 14 days of vaccination; all other adverse events were documented from the signing of the informed consent form up to approximately one month after vaccination (up to Day 43)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- 13vPnC (50 to 64 Years of Age): 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a single dose of 0.5 milliliters (mL) intramuscularly (IM) to participants 50 to 64 years of age.
  For Other Adverse Events (non-serious events): the number affected (N) for nonsystematic (unsolicited) Other Adverse Events N=80; systematic (solicited) Local Reactions N=120; systematic (solicited) Systemic Events N=112. Serious AEs were grouped by organ system, with frequency of events summarized. Non-serious AEs were summarized in a similar manner and include unsolicited AEs collected in the e-diary (systematic assessment) and solicited events collected on the case report form (non-systematic methods).
- 13vPnC (≥65 Years of Age): 13vPnC administered as a single dose of 0.5 mL IM to participants ≥65 years of age.
  For Other Adverse Events (non-serious events): the number affected (N) for nonsystematic (unsolicited) Other Adverse Events N=77; systematic (solicited) Local Reactions N=118; systematic (solicited) Systemic Events N=116. Serious AEs were grouped by organ system, with frequency of events summarized. Non-serious AEs were summarized in a similar manner and include unsolicited AEs collected in the e-diary (systematic assessment) and solicited events collected on the case report form (non-systematic methods).
Arm/Group | 13vPnC (50 to 64 Years of Age) | 13vPnC (≥65 Years of Age)
Serious Adverse Events (participants affected / at risk) | 1/134 | 1/136
Other Adverse Events (participants affected / at risk) | 120/134 | 118/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC (50 to 64 Years of Age) (N=134) | 13vPnC (≥65 Years of Age) (N=136)
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC (50 to 64 Years of Age) (N=134) | 13vPnC (≥65 Years of Age) (N=136)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 2
Dental caries (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Gingival disorder (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 0
Pericoronitis (Gastrointestinal disorders) | 1 | 0
Injection site pain (General disorders) | 53 | 52
Injection site movement impairment (General disorders) | 48 | 54
Fatigue (General disorders) | 23 | 18
Injection site erythema (General disorders) | 7 | 25
Chills (General disorders) | 6 | 8
Injection site swelling (General disorders) | 7 | 5
Pyrexia (General disorders) | 2 | 3
Axillary pain (General disorders) | 0 | 1
Feeling hot (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 10 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 16 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Redness: any (Skin and subcutaneous tissue disorders) | 7/98 | 23/110
Redness: mild (Skin and subcutaneous tissue disorders) | 7/98 | 11/110
Redness: moderate (Skin and subcutaneous tissue disorders) | 1/97 | 18/108
Redness: severe (Skin and subcutaneous tissue disorders) | 0/97 | 1/107
Swelling: any (Skin and subcutaneous tissue disorders) | 8/99 | 16/109
Swelling: mild (Skin and subcutaneous tissue disorders) | 7/98 | 8/109
Swelling: moderate (Skin and subcutaneous tissue disorders) | 2/98 | 10/108
Swelling: severe (Skin and subcutaneous tissue disorders) | 0/97 | 1/107
Pain: any (Skin and subcutaneous tissue disorders) | 60/115 | 51/115
Pain: mild (Skin and subcutaneous tissue disorders) | 56/113 | 49/115
Pain: moderate (Skin and subcutaneous tissue disorders) | 9/101 | 11/107
Pain: severe (Skin and subcutaneous tissue disorders) | 1/97 | 0/107
Limitation of arm movement: any (Skin and subcutaneous tissue disorders) | 61/115 | 63/118
Limitation of arm movement: mild (Skin and subcutaneous tissue disorders) | 59/114 | 62/118
Limitation of arm movement: moderate (Skin and subcutaneous tissue disorders) | 5/99 | 4/107
Limitation of arm movement: severe (Skin and subcutaneous tissue disorders) | 2/97 | 1/107
Fever: any ≥37.5 degrees Celsius (C) (General disorders) | 3/98 | 4/107
Fever: mild ≥37.5 degrees to <38.5 degrees C (General disorders) | 2/98 | 4/107
Fever: moderate ≥38.5 degrees to <39 degrees C (General disorders) | 1/97 | 0/107
Fatigue (General disorders) | 40/103 | 27/112
Headache (General disorders) | 26/100 | 16/111
Chills (General disorders) | 15/101 | 12/111
Rash (General disorders) | 8/98 | 14/107
Vomiting (General disorders) | 3/97 | 1/107
Decreased appetite (General disorders) | 16/99 | 10/108
New muscle pain (General disorders) | 36/105 | 33/112
Any aggravated muscle pain (General disorders) | 11/98 | 10/110
New joint pain (General disorders) | 10/100 | 13/110
Any aggravated joint pain (General disorders) | 7/98 | 6/109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.